CLINICAL TRIAL: NCT03578393
Title: Efficacy of a Preoperative Virtual Reality Intervention as a Paediatric Anxiety Improvement Strategy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Servei Central d'Anestesiologia (Other)
Responsible Party: Principal Investigator, Adriana Carbó García, Nurse, Servei Central d'Anestesiologia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRV-2017-01
Record Dates: First submitted 2018-05-30; First posted 2018-07-06 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Anxiety; Virtual Reality
Keywords: Preanesthetic visit
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Will visualize an Educational Virtual Reality video in preoperative period to reduce perioperative anxiety.
  Interventions: Device: Virtual Reality Educational Program
- Usual treatment (No Intervention): Will be applied the usual treatment (provide information on the anaesthetic-surgical process).

INTERVENTIONS:
Device: Virtual Reality Educational Program — The study group, in addition to providing the usual information about the anaesthetic-surgical process, will visualize an educational video through virtual reality glasses, of a maximum duration of 5 minutes. The video's explanation will be adapted according to the age ranges. Once the video is finished, if there aren't doubts, the visit will be concluded.
  Arms: Intervention

SUMMARY:
This study evaluate the effectiveness of the Virtual Reality Educational Program (RVEP) in the Paediatric Surgical Prehabilitation Unit to reduce the perioperative anxiety in children who undergo to elective surgery. Half of the patients will received the virtual reality program, and the other half will received de common treatment.

DETAILED DESCRIPTION:
During preoperative time, anxiety is one of the most frequent problems in children, causing an important health problem as long with pain. In the surgical fields there are two especially stressful moments for the child, the first one is the parent´s separation, and the second is the anaesthetic induction, which in up to 42% of cases can be traumatic.

Methods to treat paediatric anxiety have evolved in the last decades. Pharmacological therapy is one of the most used methods to treat anxiety in the immediate preoperative period, but complications and unwanted side effects are described. Due to this side effects, this study will evaluate the the effectiveness of the Virtual Reality Educational Program (RVEP) to reduce the perioperative anxiety in children.

ELIGIBILITY:
Inclusion Criteria:

* Children between 3 and 12 years old.
* Elective surgical intervention.
* ASA I-II (classification of the American Society of Anesthesiologists).
* Surgical complexity grade I-II according to National Institute for Clinical Excellence of the NHS.
* General anesthesia.
* Spanish or Catalan speaking families.
* Understanding the study and signing the informed consent of the study by parents or legal guardians.

Exclusion Criteria:

* Patients suffering from psychiatric or mental illness, psychomotor retardation, blindness or deafness.
* Denial of parents / legal guardians and / or children.
* Ambulatory surgery.
* Surgical intervention of the child the year before the current one.

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 241 (Actual)
Dates: Start 2019-02-02 (Actual); Primary Completion 2022-04-15 (Actual); Study Completion 2022-05-02 (Actual)

PRIMARY OUTCOMES:
Preoperative Change of Paediatric Anxiety level | 3 days: 1.- On preanesthetic visit, using mYPAS scale. 2.- The surgery day, during parents separation, using mYPAS-SF. 3.- Postoperative day (24 hours after surgery), at hospitalization room, using a mYPAS scale.
  It will be measured by modified-Yale Preoperative Anxiety Scale (mYPAS) and its short form (mYPAS-SF).
  The mYPAS score range is: 23,3 to 100, majors scores indicate anxiety. It's considerate an anxiety cut-off point scores >40, and no anxiety <40. The mYPAS-SF score range is 22,7 to 100.

SECONDARY OUTCOMES:
Paediatric pain | 2 days. The surgery day and the postoperative day (24 hours after surgery).
  Measured by Faces Pain Rating Scale o Wong Baker Faces. It consist in 6 faces, The faces represent "no harm" to "worse damage" and the score goes from 0 to 10.
Modified Aldrete postanesthetic recuperation | 1 day. The surgery day
  It is a hetero-administered scale consisting of 10 items. Each item responds to a Likert scale of 0 to 2, with a total range ranging from 0 to 10. The cut-off point is at 80% of the maximum score, ie 18 points suggest adequate recovery after anesthesia.
Parental satisfaction | 1 day. At hospital discharge (24 hours after surgery).
  Numeric Scale indicate 0= unsatisfied and 10= totally satisfied.
Resources | 1 day. The surgery day.
  Will be measured using a self-created questionnaire. It contains variables as:
  * Anaesthesia induction times (in minutes)
  * Time between the surgery ends and recovery discharge (in minutes)
  * Surgery times (in minutes)
Children's collaboration during anaesthesia induction. | 1 day. The surgery day, during anaesthesia induction.
  It will be measured by Induction Compliance Checklist (ICC). ICC score range is 0 to 10, 0 means collaborate and 10 no collaborate.
Paediatric Delirium | 2 days. The surgery day and the postoperative day (24 hours after surgery).
  Paediatric Anesthesia Emergence Delirium (PAED). It consists of 5 items with 5 possible answers on a scale of 0 to 4, with a score of > 10 indicating postsurgical agitation.

CONTACTS AND LOCATIONS:
Overall Officials: Adriana Carbó García, Nurse, Principal Investigator — Servicio Central de Anestesiología
Locations (1):
- Centro Medico Teknon, Barcelona, Spain

REFERENCES:
- [Result] Chieng YJ, Chan WC, Klainin-Yobas P, He HG. Perioperative anxiety and postoperative pain in children and adolescents undergoing elective surgical procedures: a quantitative systematic review. J Adv Nurs. 2014 Feb;70(2):243-55. doi: 10.1111/jan.12205. Epub 2013 Jul 19. PMID 23865442
- [Result] Chow CH, Van Lieshout RJ, Schmidt LA, Dobson KG, Buckley N. Systematic Review: Audiovisual Interventions for Reducing Preoperative Anxiety in Children Undergoing Elective Surgery. J Pediatr Psychol. 2016 Mar;41(2):182-203. doi: 10.1093/jpepsy/jsv094. Epub 2015 Oct 17. PMID 26476281
- [Result] Liguori S, Stacchini M, Ciofi D, Olivini N, Bisogni S, Festini F. Effectiveness of an App for Reducing Preoperative Anxiety in Children: A Randomized Clinical Trial. JAMA Pediatr. 2016 Aug 1;170(8):e160533. doi: 10.1001/jamapediatrics.2016.0533. Epub 2016 Aug 1. PMID 27294708
- [Result] Yip P, Middleton P, Cyna AM, Carlyle AV. Non-pharmacological interventions for assisting the induction of anaesthesia in children. Cochrane Database Syst Rev. 2009 Jul 8;(3):CD006447. doi: 10.1002/14651858.CD006447.pub2. PMID 19588390
- [Derived] Carbo A, Tresandi D, Tril C, Fernandez-Rodriguez D, Carrero E. Usefulness of a virtual reality educational program for reducing preoperative anxiety in children: A randomised, single-centre clinical trial. Eur J Anaesthesiol. 2024 Sep 1;41(9):657-667. doi: 10.1097/EJA.0000000000002032. Epub 2024 Jun 24. PMID 38916221